CLINICAL TRIAL: NCT06921395
Title: A Phase IV, Prospective, Randomized, Open-label, Active-controlled, Parallel-group, Multicenter Study to Evaluate Efficacy and Safety of Fang Le Shu (Recombinant FSH) Versus Guo Na Fen Used for Controlled Ovarian Stimulation in Infertile Women Undergoing In Vitro Fertilization-Embryo Transfer.
Brief Title: Phase IV Study to Evaluate the Efficacy and Safety of Fang Le Shu Compared to Guo Na Fen for Controlled Ovarian Stimulation in Infertile Women Undergoing in Vitro Fertilization-embryo Transfer (IVF-ET).
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: LG Chem (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LG-FSCL006
Record Dates: First submitted 2025-04-02; First posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Female Infertility
MeSH Terms: conditions — Infertility, Female | interventions — follitropin alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fang Le Shu (Experimental): Fang Le Shu
  Interventions: Drug: Fang Le Shu (Follitrope)
- Guo Na Fen (Active Comparator): Guo Na Fen
  Interventions: Drug: Guo Na Fen (Gonal-F)

INTERVENTIONS:
Drug: Fang Le Shu (Follitrope) — rFSH 150 IU, 225 IU, 300 IU per syringe
  Arms: Fang Le Shu
Drug: Guo Na Fen (Gonal-F) — rFSH 450 IU per pen
  Arms: Guo Na Fen

SUMMARY:
The aim of this randomized, open-label, active-controlled, parallel-group, multicenter, phase IV study is to assess the efficacy and safety of Fang Le Shu versus Guo Na Fen used for controlled ovarian stimulation in infertile women undergoing In Vitro Fertilization-Embryo Transfer.

ELIGIBILITY:
Inclusion Criteria:

* Is pre-menopausal female aged ≥20 to <40 years.
* Has regular menstrual cycles of ≥25 to ≤35 days.
* Has Normal baseline serum FSH, LH, E2, P4.
* Is able to voluntarily sign the informed consent form (ICF).
* Has history of infertility for at least 1 year before the day of randomization; however, subjects with confirmed diagnosis of infertility are eligible without fulfilling the 1-year requirement.

Exclusion Criteria:

* Has any known clinically significant major systemic disease, or endocrine or metabolic abnormalities with the exception of controlled thyroid function disease.
* Has body mass index (BMI) of >30 kg/m2.
* Has clinically significant abnormalities of the uterus, ovary, or appendix prior to the day of randomization
* Has history of surgeries that may affect oocyte retrieval or pregnancy outcome, such as surgical resection of uterine mediastinum, fibroids, or cysts (however, patients who received polypectomy are allowed to enroll).
* Has history of severe ovarian hyperstimulation syndrome (OHSS) defined as Grade 4 or higher.
* Poor ovarian reponder according to Bologna criteria
* Has plans to donate oocyte or recieve embryo from another women or undergo preimplantation genetic testing(PGT)
* Has history of three or more failures in previous IVF cycles
* Has history of recurrent miscarriage
* Has known current active pelvic inflammatory disease.
* Is currently breastfeeding.
* Has a contraindication to pregnancy that would preclude participation in the trial.

Ages: 20 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 248 (Estimated)
Dates: Start 2025-02-15 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of oocytes retrieved | 36 ± 3 hours after HGC trigger

SECONDARY OUTCOMES:
High quality embryo rate | 3 days after oocyte retrieval
Biochemical pregnancy rate | 14 days after embryo transfer
Clinical pregnancy rate | 5 weeks after embryo transfer
Ongoing pregnancy rate | 10 weeks after embryo transfer
Miscarriage rate | 28 weeks of gestation
Live birth rate | 40 weeks of gestation

CONTACTS AND LOCATIONS:
Locations (1):
- The first affiliated hospital of Zhengzhou University, Zhengzhou, China

IPD SHARING:
Plan to Share IPD: No